CLINICAL TRIAL: NCT05331716
Title: Substrate Based Modification in Ventricular Tachycardia: Ablation of the Local Abnormal Ventricular Activity Only
Brief Title: Modification of the Local Abnormal Ventricular Activity Only
Acronym: LAVAONLY
Status: Completed | Type: Observational
Sponsor: University of Kiel (Other)
Collaborators: Krankenhaus Landshut Achdorf (Unknown)
Responsible Party: Principal Investigator, Prof. Dr. Hendrik Bonnemeier, Coordinating principal investigator, University of Kiel
Other Study IDs: 2021-1232
Record Dates: First submitted 2022-04-04; First posted 2022-04-18 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Ventricular Tachycardia
Keywords: local abnormal ventricular activity; substrate modification; electrophysiology; LAVA; decremental
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Cardiac ablation therapy — In a subset of patients with known therapy refractory arrhythmia sole LAVA modification is fashioned
  Other Names: LAVA modification

SUMMARY:
Local abnormal ventricular activity (LAVA) is composed of high-frequency, mainly low voltage signals that represent near-field signals from slow-conducting tissue and thus potential VT isthmuses. The identification of LAVA potentials and their modification have usually been a complimentary component of the substrate-based modification of scar related ventricular arrhtyhmias. With better identification through technical solutions and improved algorithms, LAVA modification may be feasible for treatment in therapy refractory VT.

DETAILED DESCRIPTION:
As of 2019 we started LAVA modification only in a subset of patients with therapy refractory ventricular tachycardia. The cohort icludes 55% patient with ischemic cardiomyopathy and 45% with dilated cardiomyopathy. 80% are ICD recipients. These patients were now retrospectively analysed in depth. The endpoint is time to relapse of ventricular tachycardia or ICD shock or death due to malignant arrhythmia. We evaluated all patients we treated accordingly from March 2019 through October 2020. No patient was excluded.

ELIGIBILITY:
Inclusion Criteria:

therapy refractory ventricular arrhythmia

Exclusion Criteria:

none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all consecutive patients undergone LAVA modification alone for treatment of therapy refractory ventricular arrhythmia
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
VT | 12 months
  occurrence/documentation of ventricular arrhythmia in participant after substrate modification during follow-up period (either Holter ECG or defibrillator interogation or ILR/ICM or electrophysiology study)
appropriate therapy delivered by defibrillator (ICD) | 12 months
  appropriate therapy (shock, ATP) delivered by ICD in participants during follow-up period
death | 12 months
  patient succumbed due to malignant ventricular arrhythmia or therapy

SECONDARY OUTCOMES:
death any cause | 36 months
  death any cause during observation period

CONTACTS AND LOCATIONS:
Overall Officials: Hendrik Bonnemeier, PhD, Study Director — University of Kiel - Medical Faculty; Stefan Borov, MD, Principal Investigator — University of Kiel - Medical Faculty
Locations (1):
- Krankenhaus Landshut Achdorf, Landshut, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Yes
Spreadsheet with characteristics (e.g.; procedure time, etc)
Supporting Information: Study Protocol